CLINICAL TRIAL: NCT04342533
Title: Prospective Randomized Trial of Irritative Symptoms Severity Assessment After Holmium Laser Enucleation of the Prostate (HoLEP) Versus Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP).
Brief Title: Prospective Randomized Trial of Irritative Symptoms Severity Assessment After (HoLEP) Versus ThuFLEP
Acronym: PRISSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy director for research, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sechenov-Ho_Vs_TFL-20
Record Dates: First submitted 2020-03-12; First posted 2020-04-13 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: BPH; Prostate Obstruction
Keywords: HoLEP; ThuFLEP; EEP; prostate enucleation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ThuFLEP (Experimental): Patients who underwent thulium fiber enucleation of the prostate
  Interventions: Procedure: Thulium fiber laser enucleation of the prostate
- HoLEP (Active Comparator): Patients who underwent holmium laser enucleation of the prostate
  Interventions: Procedure: Holmium laser enucleation of the prostate

INTERVENTIONS:
Procedure: Thulium fiber laser enucleation of the prostate — enucleation of the BPH according to standard procedure protocol
  Other Names: ThuFLEP
  Arms: ThuFLEP
Procedure: Holmium laser enucleation of the prostate — enucleation of the BPH according to standard procedure protocol
  Other Names: HoLEP
  Arms: HoLEP

SUMMARY:
The investigators hypothesize that the functional outcomes of both techniques are comparable. However, ThuFLEP might increase speed recovery of postoperative irritation and early stress urinary incontinence according to the Questionnaire for Urinary Incontinence Diagnosis (QUID) because of minimal tissue penetration depth of TFL.

DETAILED DESCRIPTION:
Thulium fiber laser enucleation of the prostate (ThuFLEP) has already shown the outcomes comparable to OSP with better safety profile (lower blood loss compared to OSP) and shorter hospital stay. TFL has the efficacy and safety proven in comparative trials, being a promising rival for HoLEP. The main features of TFL distinguishing it from Ho:YAG is its wavelength of 1.94 µm (leading to about three-fold increase in water absorption and lesser penetration depth of <0.1 mm vs >0.2 mm in Ho:YAG). With identical average and peak powers of 100 W, the laser does not burst tissues, allowing for clean and precise cutting instead. Conversely, Ho:YAG's average power is about 100 W and its presumable peak power is around 10-15 kW. With such an outburst of energy, each pulse of Ho:YAG creates a large vapor bubble which ruptures the tissue. This may be a possible reason for increased irritative symptoms in early postoperative period after HoLEP comparing to ThuFLEP. But all in all, the probable causes for such postoperative symptoms remain unclear so far, despite the fact that absence of irritation and incontinence is ought to be one quality marker of "Pentafecta". According to the idea of high-power impact, probably, decreasing of HoLEP power will mitigate these problems. On the one hand, low-power HoLEP is feasible, safe and effective modality for symptomatic BPO. However, the results remain controversial and there is lack of LP-HoLEP application data nowadays. May be, with another option, for instance OSP or monopolar enucleation, it is possible to solve the issues. But the discussion of the past years demonstrates that the presence of early SUI is not only a problem of EEP, but also underreported in other approaches in relieving BPO secondary to BPH.

ELIGIBILITY:
Inclusion Criteria:

* LUTS presence, proven by:

  1. IPSS questionnaire (Score >20);
  2. OR uroflowmetry result (Qmax <10 ml/s);

Exclusion Criteria:

* Prostate volume > 120 cc
* Prostate cancer on pathology;
* Urethral strictures;
* Bladder calculi;
* Prior prostate surgery;
* Neurogenic bladder dysfunction.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — presence of prostate and BPH
Enrollment: 140 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
severity of urinary incontinence | change from 1 week to 6 months after surgery
  Questionnaire for Urinary Incontinence Diagnosis (higher score means worse incontinence)

SECONDARY OUTCOMES:
rate of intra- and perioperative adverse events | 6 months follow up
  complications according to Clavien-Dindo classification (higher score means more severe complication)
surgery duration | during surgery
  lengths of the procedure
hemoglobin drop | 1 day after surgery
  decrease of hemoglobin at the first day after surgery comparing to preoperative value
catheter stay | 1 week after surgery
  lengths of catheterization
hospitalization length | 1 week after surgery
  duration of staying at hospital after the surgery
functional outcomes | change from 3 to 6 months after surgery
  IPSS (international prostate symptos score), QoL (quality of life), IIEF-5 (international index of erectile function) questionaries, Qmax

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No